CLINICAL TRIAL: NCT00724243
Title: Remicade Treatment Registry in Rheumatoid Arthritis I
Brief Title: Safety and Effectiveness of Infliximab in Slovakia When Used for Rheumatoid Arthritis (Study P04741)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04741
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2010-02-19 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis Patients in Slovakia: Rheumatoid arthritis patients in Slovakia who are starting treatment with infliximab for the first time, in accordance with normal clinical practice.
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab given in accordance with the local summary of product characteristics
  Other Names: Remicade; SCH 215596

SUMMARY:
This study will gather information on the safety and efficacy of patients with rheumatoid arthritis (RA) who are starting treatment with infliximab for the first time. Patients will be treated in the usual manner according to local guidelines and normal clinical practice.

DETAILED DESCRIPTION:
Local patients, diagnosed with RA at the National Institute of Rheumatic Diseases, Piestany, Slovakia, can participate, if their physicians have decided to treat the patient with infliximab. Registration for the trial will be done on a voluntary basis.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have been given patient leaflet,
* Subject must not have ever received infliximab at the time of registration,
* Subject must be a good candidate for infliximab as per Summary of Product Characteristics
* Subject must sign the approved consent form

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects for this study will be patients expecting to initiate infliximab, for the first time, for the diagnoses of rheumatoid arthritis at the National Institute of Rheumatology Diseases in Piestany, Slovakia.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2006-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Infliximab: Rheumatoid arthritis patients in Slovakia who are starting treatment with infliximab for the first time, in accordance with normal clinical practice.
Period: Overall Study
Arm/Group | Infliximab
Started | 33
Completed | 18
Not Completed | 15
Not completed — Lack of Efficacy | 10
Not completed — Adverse Event | 5

BASELINE CHARACTERISTICS:
Arm/Group | Infliximab
Number analyzed (Participants) | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.38 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 7
Region of Enrollment [Number; unit: participants]
  Slovakia | 33

OUTCOME MEASURES:

1. Primary Outcome: Average Change in Disease Activity Score 28 (DAS 28) From the Beginning of the Treatment
Description: The DAS 28 is an assessment of disease activity based on swollen joint count, erythrocyte sedimentation rate, and general health. Participants can be scored on a range of 0 to 10, with lower scores indicating less disease activity.
Time Frame: Baseline, Week 14, and Week 54
Population: Thirty-three participants had a DAS 28 score at the beginning of treatment.
  Twenty-eight participants had a DAS 28 score at Week 14.
  Twenty-two participants had a DAS 28 score at Week 54.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Infliximab
Number analyzed (Participants) | 33
Units on a Scale
  Baseline | 7.11 (0.65)
  Week 14 | 2.94 (1.22)
  Week 54 | 3.27 (1.59)

2. Primary Outcome: Number of Participants Fulfilling Criteria for a Therapeutic Response According to the European League Against Rheumatism (EULAR) Response Criteria
Description: Response to treatment was assessed by EULAR response criteria. According to these criteria, participants were characterized as good, moderate, or non-responders based on both DAS level attained and change in DAS. Good response was defined as >1.2 improvement in DAS from Baseline and DAS attained during follow-up of ≤2.4. Non-responders were participants with improvement of ≤0.6 or participants with improvement of >0.6 but ≤1.2 and DAS attained during follow-up of >3.7. Remaining participants were classified as moderate. Scores of good and moderate were considered to have therapeutic response.
Time Frame: Week 14 and Week 54
Measure: Number; unit: Participants
Arm/Group | Infliximab
Number analyzed (Participants) | 33
Participants
  Week 14 | 27
  Week 54 | 19

ADVERSE EVENTS:
Arm/Group | Infliximab
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 4/33
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab (N=33)
Allergic reactions to infusion (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contractor agrees to acknowledge his contractual relationship with Sponsor in his lecturing or publication activities in relation to subject matter and/or in relation to any other matter concerning Sponsor. However, unless Sponsor's prior consent was given, Contractor shall not specify in more detail the content or subject matter of his contract. Contractor shall not publish or provide to 3rd parties for publication purposes any results of his activities without Sponsor's prior written consent.